CLINICAL TRIAL: NCT06055296
Title: Multisite Implementation of COMPRENDO (ChildhOod Malignancy Peer REsearch NavigatiOn) to Improve Participation of Hispanic Children in Cancer Clinical Trials
Brief Title: Multisite Implementation of COMPRENDO
Acronym: COMPRENDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of California, San Francisco (Other); University of Alabama at Birmingham (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, M. Paula Aristizabal, Associate Professor of Clinical Pediatrics, Division of Pediatric Hematology/Oncology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 808092; 1R01CA279945-01 (NIH)
Record Dates: First submitted 2023-09-01; First posted 2023-09-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: Research Literacy; Cancer Disparities; Minority Clinical Trial Accrual; Patient Navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: We will use a Hybrid 1 design that combines a randomized effectiveness trial and a mixed methods observational implementation evaluation. Hybrid designs assess both clinical effectiveness and implementation, thus bridging the gap between two research areas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPRENDO Intervention (Experimental): Parent participants randomized to the intervention group will receive the COMPRENDO intervention that includes 2-4 visits led by a peer navigator across a 4-week period. Navigator visits will last about 16 - 60 minutes depending upon the needs and desires of the parent. Navigator sessions will be conducted in the parents' preferred language (either English or Spanish). Peer navigators will:
  * Discuss general concepts related to informed consent and treatment options, including standard of care and clinical trials. The navigator will not discuss specific medications with parents.
  * Attend the informed consent discussion parents have with their child's oncologist.
  * Help parents come up with questions when the oncologist talks about cancer treatment options.
  * Go over the consent forms. Answer questions parents may have to the best of their ability.
  * Meet with parents over 4 weeks. During these meetings, the navigator will facilitate decision-making.
  Interventions: Other: COMPRENDO Peer Navigation Intervention
- Usual Care (No Intervention): Parents will participate in an informed consent conference with the oncologist to discuss treatment options for the child as per each institution's procedure.

INTERVENTIONS:
Other: COMPRENDO Peer Navigation Intervention — Parents randomized to the intervention, COMPRENDO, will receive culture, language, and health literacy-concordant pre-accrual, accrual, and post-accrual activities in person led by a peer navigator for up to 4 weeks. Visit 1 (V1) will provide anticipatory guidance and education on a) general concepts of pediatric cancer research (standard of care, clinical trials, randomization); b) informed consent/assent, research affiliations (e.g., Children's Oncology Group); c) clinical trial types (therapeutic, non-therapeutic); d) voluntariness; and e) "frequently asked questions", resources. Navigators will follow a script supported by culture, language and health-literacy concordant handouts and graphic materials, decision aids, and short video-clips. Navigators also provide support with decision-making and answer parents' questions. Three follow-up peer navigator visits (V2, V3, V4) over 4 weeks are tailored to the parents' needs.
  Arms: COMPRENDO Intervention

SUMMARY:
COMPRENDO (ChildhOod Malignancy Peer Research NavigatiOn) is a multi-site randomized clinical trial (RCT) that uses a Hybrid Type 1 design, to test the effects of a clinical intervention on patient-level outcomes, while exploring multilevel implementation factors that can inform real-world setting implementation. This study will test the impact of COMPRENDO, a peer-navigation intervention, vs. usual care on accrual to childhood cancer therapeutic clinical trials and parental informed consent outcomes. COMPRENDO will be delivered by trained peer navigators in 4 visits. A mixed methods (surveys, individual interviews) implementation evaluation will examine implementation factors that can inform the use of peer navigation in clinical practice, integrating data from clinicians, navigators, administrators, and parents pre and post the RCT.

DETAILED DESCRIPTION:
Aim 1:

Test the effectiveness of COMPRENDO vs. usual care to increase clinical trial accrual in a multisite RCT.

Aim 2:

Determine the impact of COMPRENDO vs. usual care on parental outcomes (informed consent, comprehension, voluntariness, decision-making self-efficacy, satisfaction with informed consent and decisional regret).

Aim 3:

Evaluate multisite implementation of COMPRENDO, focusing on acceptability, feasibility, and fidelity. We will use mixed methods with a minimum of 50 stakeholders: 22 clinicians, (17 oncologists, 3 psychologists, 2 social workers), 4 navigators, 4 administrators and 20 parents to identify implementation factors.

Within each site, eligible participants will be randomized 1:1 to the intervention vs. usual care (informed consent discussion with the oncologist only), resulting in ≈200 participants randomized to each arm.

ELIGIBILITY:
Participants (n≈400) will be parents of Hispanic children (0-17 years) with newly diagnosed cancer or cancer-like disease (histiocytic disorders or myelodysplastic syndromes) and eligible for a therapeutic clinical trial who meet the following inclusion criteria:

* are a Hispanic parent/primary legal guardian;
* has a child aged 0 to 17 y with a new diagnosis of cancer or cancer-like disease (histiocytic disorders or myelodysplastic syndromes);
* has a child who is eligible for a therapeutic cancer clinical trial;
* will participate in an informed consent discussion for the therapeutic clinical trial;
* has an understanding of written and spoken English or Spanish;
* has signed the consent form for the proposed COMPRENDO study.

Parent Exclusion Criteria:

* second malignancy/relapse;
* diagnosed at an outside institution;
* potential transfer of care to another institution within the next 4 months;
* previously on a clinical trial;
* does not understand written and spoken English or Spanish;
* not Hispanic.

Stakeholder Inclusion Criteria:

Clinicians and parents of children with cancer who have participated in IC discussion for a cancer therapeutic clinical trial.

Stakeholder Exclusion Criteria:

Clinicians and parents of children with cancer who have not participated in IC discussion for a cancer therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Accrual | 12 weeks
  Measured by a higher proportion of children enrolled in therapeutic trials whose parents are randomized to COMPRENDO vs. the proportion of children enrolled in therapeutic trials whose parents are randomized to usual care.

SECONDARY OUTCOMES:
Informed Consent Comprehension | 12 weeks
  Informed Consent Comprehension will be assessed using the Quality of Informed Consent (QuIC), a valid 20-item instrument that assesses objective understanding of the basic elements of Informed Consent. The summary score potentially ranges from 0 to 100. The highest the summary score, the highest the comprehension.
Voluntariness | 12 weeks
  Voluntariness will be assessed using the Decision-making Control Instrument (DMCI), a 9-item, Likert-format scale, which is used in parents who make decisions about research, including cancer. The instrument score range from 9-54, the higher score equals to higher perception of voluntariness.
Decision-Making Self-Efficacy | 12 weeks
  Decision-Making Self Efficacy will be assessed with the 11-item Decision Self-Efficacy Scale (DSE), a 5-point scale which measures self-confidence in decision making (shared decision making, decision conflict, feeling informed and supported). Score range from 0 [not at all confident] to 100 [very confident]. A score of 0 means extremely low self efficacy and a score of 100 means extremely high self efficacy.
Decisional Regret | 12 weeks
  The 5-item Decisional Regret Scale will measure regret after health-care decisions. Score range is from 0 to 100. A score of 0 means no regret; a score of 100 means high regret.
Satisfaction with informed consent | 12 weeks
  Satisfaction with informed consent will be measured with a 24-item satisfaction questionnaire to evaluate parents' perceptions of overall satisfaction with the IC discussion (satisfaction with ICs explanation, quantity of information, utility of the IC, affective responses).The score ranges from 7-21. A score of 7 meaning least satisfied; a score of 21 most satisfied.
Trust in Research | 12 Weeks
  Assesses individual's views on research studies.

OTHER OUTCOMES:
Acceptability (parents) | Year 1-Year 5
  Acceptability of COMPRENDO will be assessed in parents the 9-item Patient Satisfaction with Navigator (PSN-I). The score ranges from 9-45. A higher score on the PSN-I indicates higher satisfaction with their interpersonal relationship with the patient navigator. Our acceptability goal is >80%
Acceptability (clinicians) | Year 1-Year 5
  Acceptability of COMPRENDO will be assessed in clinicians with the 6-item Intervention Credibility Scale. The score ranges from 4-20. Higher scores indicate greater acceptability. Our acceptability goal is >80%
Feasibility | Year 1-Year 5
  Feasibility will be assessed by 4-item Feasibility of Intervention measure. The score ranges from 4-20. Higher scores indicate greater feasibility. Our feasibility goal is >80%.
Fidelity | Year 1-Year 5
  Fidelity will be assessed by measuring adherence to the fidelity navigator checklist. Our fidelity goal is >90%.

CONTACTS AND LOCATIONS:
Overall Officials: M.Paula Aristizabal, MD, MAS, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - Children's of Alabama/University of Alabama at Birmingham, Birmingham, Alabama
  - Rady Children's Hospital San Diego/University of California San Diego Moores Cancer Center, San Diego, California
  - University of California San Francisco Benioff Children's Hospitals, San Francisco, California
  - Dana Farber Cancer Institute/Boston Children's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Palinkas LA, Mendon SJ, Hamilton AB. Innovations in Mixed Methods Evaluations. Annu Rev Public Health. 2019 Apr 1;40:423-442. doi: 10.1146/annurev-publhealth-040218-044215. Epub 2019 Jan 11. PMID 30633710
- [Background] Moullin JC, Dickson KS, Stadnick NA, Rabin B, Aarons GA. Systematic review of the Exploration, Preparation, Implementation, Sustainment (EPIS) framework. Implement Sci. 2019 Jan 5;14(1):1. doi: 10.1186/s13012-018-0842-6. PMID 30611302
- [Background] Freeman HP. Patient navigation: a community based strategy to reduce cancer disparities. J Urban Health. 2006 Mar;83(2):139-41. doi: 10.1007/s11524-006-9030-0. No abstract available. PMID 16736361